CLINICAL TRIAL: NCT07153354
Title: Precision of Patient-specific Screw Holes Locating Surgical Guide and Pre-bent Plates Osteosynthesis Versus Classical Workflow in the Management of Class IV Mandibular Fractures
Brief Title: Patient-Specific Guides vs. Classical Workflow in Class IV Mandibular Fracture Fixation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed abdelsalam Gaber elkhouly (Other)
Responsible Party: Sponsor-Investigator, Mohamed abdelsalam Gaber elkhouly, Resident oral and maxillo-facial surgery, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3D-T4F-RCT-2025
Record Dates: First submitted 2025-05-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Mandibular Class Iv Fractures
Keywords: Per-bent plates; Class iv mandibular fractures; Surgical guide; patient-specific screw holes locating surgical guide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient-specific screw holes locating surgical guide and pre-bent plates osteosynthesis (Experimental): Patients In this group will be reduced using patient computer-guided specific screw holes locating guide and pre-bent plates(2.3 for inferior border and 2.0 for superior border)
  Interventions: Device: patient-specific screw holes locating surgical guide and pre-bent plates
- classical work-flow (Active Comparator): Patients In this group will be reduced by classical reduction and fixation protocol
  Interventions: Device: 2 titanium per-bent mini plates

INTERVENTIONS:
Device: patient-specific screw holes locating surgical guide and pre-bent plates — Virtual reduction of the fracture will be done, followed by 3D printing of the corrected mandible model. Plates will be pre-bent on the model, then scanned in position to create a surgical guide for accurate screw hole placement during surgery.
  Arms: patient-specific screw holes locating surgical guide and pre-bent plates osteosynthesis
Device: 2 titanium per-bent mini plates — The fixation will be performed according to established surgical principles for managing class iv mandibular fractures, without patient-specific planning
  Arms: classical work-flow

SUMMARY:
This study aims to overcome the limitations of current, standard approach of mandibular fracture reduction and fixation including improper alignment of segments, malocclusion, nerve affections and related teeth roots injury. The introduction of Computer Aided designing/Computer Aided manufacturing software has provided surgeons with an opportunity to perform virtual manipulations of computed tomography datasets preoperatively and production of corrected mandibular model for plate pre-bending and fabrication of plate locating surgical guide which provide accurate segment reduction and fixation with accurate post-operative occlusion and minimal post-operative complication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with delayed mandibular class IV fracture need open reduction and internal fixation.
* Patients with a medical history that did not hinder plate placement (uncontrolled diabetes) and adequate proper oral hygiene.
* Both genders, males and females, will be included

Exclusion Criteria:

* General contraindications to surgery.
* Patients with unfavorable or comminuted fractures.
* Subjected to irradiation in the head and neck area less than 1 year before fixation.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Patients participating in other studies, if the present protocol could not be properly followed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of fracture reduction | Within one week postoperatively
  Accuracy of fracture reduction, measured as the mean linear deviation (in millimeters) between the postoperative Computed Tomography scan and the preoperative virtual surgical plan
  Method of assessment: Postoperative Computed Tomography scans will be superimposed onto the preoperative virtual plan using 3D analysis software (e.g., Mimics/3-matic or equivalent). Linear and angular deviations of fracture segments will be calculated at predefined anatomical landmarks.

SECONDARY OUTCOMES:
Occlusion | At 1 week, 1 month, 3 months, and 6 months postoperatively
  change in occlusion will be assessed by a maxillofacial surgeon at each follow-up visit (1 week, 1 month, 3 months, 6 months postoperatively) using Angle's classification and clinical examination.
  Unit of Measure: Presence/absence of malocclusion (Yes/No)
Operation time | During the surgery
  Total duration from skin incision to wound closure, recorded intraoperatively.